CLINICAL TRIAL: NCT06493266
Title: The Effect of Neurolingualistik Programming (NLP) on Pain Score, Fear of Pain and Pain Catastrophizing Before Colposcopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Alev Esercan, MD, Sanliurfa Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 63-seah 2
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Pain, Acute
Keywords: pain; NLP; colposcopy
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): pain evaluation by questionnaire in colposcopy patients
- intervention (Experimental): pain evaluation by questionnaire in colposcopy patients after NLP
  Interventions: Behavioral: neurolinguistic programmino

INTERVENTIONS:
Behavioral: neurolinguistic programmino — In this randomized controlled study, the group of patients with an indication for colposcopy in the Gynecological Oncology Department of Şanlıurfa Training and Research Hospital, Department of Gynecology and Obstetrics, will be divided into two groups and NLP training will be given before colposcopy in a double-blind manner, and after colposcopy, VAS (visual pain scale), fear of pain scale will be given. 3, evaluation will be made using the pain catastrophizing scale. NLP training will be given for approximately 20 minutes, and the group that will not receive NLP training will remain silent for 20 minutes. The results will be compared.
  Arms: intervention

SUMMARY:
Colposcopy, evaluation of cervical cytological abnormalities and It is the gold standard procedure for the early diagnosis of preinvasive and invasive diseases. Despite her Essentially a minimally invasive intervention, even referring the patient to colposcopy can cause significant anxiety and distress in patients. Increased anxiety can also lead to deterioration in health-related quality. Studies have been conducted to reduce the anxiety of women undergoing colposcopy, but there are no publications on topics such as anxiety, pain perception, and pain catastrophizing.

Neuro Linguistic Programming (NLP) has been called "the art and science of personal excellence", "the study of subjective experience". NLP helps us understand the difference between our actions that produce mediocre results or failure and those that require success or excellence.

NLP: "How do I do something I do well?", "How can I do it better?", "How can I gain skills that I admire in others? It addresses questions like ". It is important to note that NLP is not limited to observable behavior. Our way of thinking, that is, all experience and It also includes the mental processes that control our actions. By dealing with the entire structure of a person's experience (in fact, their motivation), it tries to shape the thought processes, emotions and beliefs that result in a behavior. It is especially about our communication with ourselves as well as with others.

No study was planned on pain and pain perception during colposcopy by teaching the NLP technique to the patients.

ELIGIBILITY:
Inclusion Criteria:Those who are over 18 years of age and are not pregnant with an indication for colposcopy; Those who agreed to participate in the study,

Exclusion Criteria:patients who understand and can speak Turkish patients who did not meet the inclusion criteria or had previously undergone colposcopy - -

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — colposcpoy patients
Enrollment: 100 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
pain evaluation | 1 hour
  pain level

CONTACTS AND LOCATIONS:
Overall Officials: aysegül kılıçlı, Study Chair — Sanliurfa Education and Research Hospital
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 months